CLINICAL TRIAL: NCT02009033
Title: Effect of Colloid Versus Crystalloid on Coagulation in Elective Urological Surgery. A Randomised Clinical Study
Brief Title: Effect of Colloid Versus Crystalloid on Coagulation in Elective Urological Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: K. C. Rasmussen (Other)
Responsible Party: Sponsor-Investigator, K. C. Rasmussen, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-2-2011-063
Record Dates: First submitted 2011-07-18; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Disorders of Coagulation
MeSH Terms: conditions — Hemostatic Disorders | interventions — Ringer's Lactate; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ringer's lactate (Experimental): Fluid therapy during operation
  Interventions: Drug: Lactated Ringer; Drug: Hydroxyethylstarch

INTERVENTIONS:
Drug: Lactated Ringer — When normovolæmic status of the patient is secured, 35 ml/kg of the allocated fluid is infused during the operation (estimated time for this type of operation is 180 minutes), however max. 3500 ml.Lactated Ringer is the interventional medication.
Drug: Hydroxyethylstarch

SUMMARY:
The purpose of this study is to investigate the effect of thin fluid with starch versus thin fluid without starch on coagulation in elective surgery when the patient is normovolæmic during operation.

DETAILED DESCRIPTION:
The primary goal is to register coagulation on basis of blood samples inclusive thromboelastography results.

The secondary goal is to register blood loss and use of blood products during operation.

The trial concerns 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years.
* Indication for elective surgery with removal of the urine bladder.
* Patient without anticoagulative, acethylsalisylsyre or NSAID medicine during the last 5 days,if using.

Exclusion Criteria:

* Cerebral haemorrhage
* Renal insufficiency demanding dialysis
* Manifest cardiac and hepatic insufficiency
* Disturbance in coagulation
* Hypernatriæmi
* Hyperchloræmi
* Pregnant or nursing
* Allergic to hydroxyethylstarch
* Participating in another trial-if interferring the present trial
* Incapable of managing his own affairs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Estimate coagulation on basis of bloodsamples | 6 months

SECONDARY OUTCOMES:
Estimate coagulation by bloodloss and need for transfusion | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Niels Henry Secher, Professor, Study Chair — Rigshospitalet , Dept. 2042, 2100 Copenhagen